CLINICAL TRIAL: NCT04717310
Title: A Randomized, Double-blind, Vehicle-Controlled, Seamless and Adaptive-designed Phase II/III Study to Evaluate the Efficacy and Safety of Topical SHR0302 Ointment in Adult Patients With Mild-to-Moderate Atopic Dermatitis
Brief Title: Evaluate the Efficacy and Safety of Topical SHR0302 Ointment in Patients With Mild-to-Moderate Atopic Dermatitis
Acronym: MARBLE-23
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Reistone Biopharma Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RSJ10431
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Active Comparator: SHR0302 Ointment Dose#1 (Active Comparator): Drug: SHR0302 Ointment Twice a day (BID)
  Interventions: Drug: SHR0302 Ointment
- Active Comparator: SHR0302 Ointment Dose#2 (Active Comparator): Drug: SHR0302 Ointment Twice a day (BID)
  Interventions: Drug: SHR0302 Ointment
- Active Comparator: SHR0302 Ointment Dose#3 (Active Comparator): Drug: SHR0302 Ointment Twice a day (BID)
  Interventions: Drug: SHR0302 Ointment
- Placebo Comparator: Placebo (Placebo Comparator): Drug: Vehicle Twice a day (BID)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: SHR0302 Ointment — SHR0302 Ointment Twice a day (BID)
  Other Names: SHR0302 Ointment 2%
  Arms: Active Comparator: SHR0302 Ointment Dose#1
Drug: SHR0302 Ointment — SHR0302 Ointment Twice a day (BID)
  Other Names: SHR0302 Ointment 1%
  Arms: Active Comparator: SHR0302 Ointment Dose#2
Drug: SHR0302 Ointment — SHR0302 Ointment Twice a day (BID)
  Other Names: SHR0302 Ointment 0.5%
  Arms: Active Comparator: SHR0302 Ointment Dose#3
Drug: Vehicle — Twice a day (BID)
  Other Names: Placebo
  Arms: Placebo Comparator: Placebo

SUMMARY:
This is a Randomized, Double-blind, Vehicle-Controlled, Seamless and Adaptive-designed Phase II/III Study to Evaluate the Efficacy and Safety of Topical SHR0302 Ointment in Adult Patients with Mild-to-Moderate Atopic Dermatitis.

It will consist of phase II and phase III parts, phase II will be a dose-ranging part and phase III will be a pivotal study part.

DETAILED DESCRIPTION:
This study will evaluate the topical SHR0302 ointment, a JAK (Janus Kinase) inhibitor, in atopic dermatitis patients. The EASI (Eczema Area and Severity Index), IGA (immunoglobulin A), SCORAD (Scoring of Atopic Dermatitis),DLQI (Dermatology Life Quality Index)and NRS (Numeric Rating Score) will be applied to assesses to the efficacy, and other safety measurements will be also collected within the whole study duration.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject at least at ≥18 and ≤75years of age at time of informed consent.
* Have mild-to- moderate AD (Atopic Dermatitis), as determined by all of the following:

  1. Were diagnosed with AD (defined by the Hanifin and Rajka criteria)
  2. With AD history at least 6 months
* Capable of providing a signed and dated informed consent form indicating the subject has been informed of all pertinent aspect of the study
* All women of childbearing potential and all men must be willing to use at least one highly effective method of contraception from signing of informed consent, throughout the duration of the study, and for 28 days after last dose of study medication.

Exclusion Criteria:

* Subjects currently have active forms of other skin disease (e.g., psoriasis, or lupus erythematosus) that would interfere with evaluation of the effect of study medication on atopic dermatitis, or skin infections (bacteria, fungi, or viruses), or diseases that can cause skin itching (such as itching caused by diabetes), or subjects who are allergic to topical skin drugs
* Subjects with serious concomitant illness that could require administering of systemic corticosteroids or otherwise interfere with study participation or require active frequent monitoring (e.g. unstable chronic asthma)
* Subjects who have a history of mental illness or disease such as anxiety and depression, and are not suitable to participate in this study
* Subjects with serious and uncontrolled disease that may affect the safety of the subject, compliance, affect the evaluation of the endpoint, or require the use of drugs that are not allowed in the protocol
* Subjects with Human immunodeficiency virus (HIV), or hepatitis B virus ,or hepatitis C virus ,or syphilis related laboratory test positive (subjects positive for hepatitis B surface antigen, HBV (hepatitis B virus) DNA must be greater than lower limit of detection
* Subjects with malignant tumors or a history of malignant tumors, except for fully treated or resected skin non-metastatic basal cell carcinoma or squamous cell carcinoma
* Pregnant female subjects, breastfeeding female subjects, or male subjects able to father children and female subjects of childbearing potential who are unwilling or unable to use a highly effective method of contraception as outlined in protocol for the duration of the study and for at least 28 days after last dose of investigational product.
* The investigators determined that there were conditions that affected the safety and efficacy of the investigational drug
* Subjects who, in the opinion of the investigator or Reistone, will be unsuitable for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 645 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2023-09-08 (Estimated); Study Completion 2024-07-14 (Estimated)

PRIMARY OUTCOMES:
Percentage change from baseline in the eczema area and severity index (EASI) total score at Week 8 | 8 weeks
  The percentage of subjects achieving the Investigator's Global Assessment（IGA）of clear (0) or almost clear (1) with a ≥2 points improvement from baseline at Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Yanhong Cheng, Study Director — Reistone Pharma
Locations (31):
- China (31):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - The First Hospital Affiliated to AMU (Southwest Hospital), Chongqing, Chongqing Municipality
  - Xinqiao Hospital of AMU, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Nanyang first people's Hospital, Nanyang, Henan
  - Wuhan NO.1 Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second People's Hospital of Wuxi, Wuxi, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jiangxi Provincial Hospital of Dermatology, Nanchang, Jiangxi
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - SIR RUN RUN Shaw Hospital Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Hangzhou Third People's Hospital, Hangzhou, Zhejiang
  - Hwa Mei Hospital, Ningbo, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The Third Xiangya Hospital of Central South University, Changsha
  - Sun. Yat- Sen Memorial Hospital, Sun. Yat- Sen University, Guangzhou
  - Zhejiang province People's Hospital, Hangzhou
  - Huashan Hospital Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No